CLINICAL TRIAL: NCT00205244
Title: Preoperative Preparation for Children: Use of Relaxation and Distraction
Brief Title: Preoperative Preparation for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2003-0495
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Elective Surgery; Anxiety
MeSH Terms: conditions — Anxiety Disorders

INTERVENTIONS:
Behavioral: Healing images, relaxation and distraction materials

SUMMARY:
Children scheduled for elective surgery are randomized into a control and intervention group. Children in the intervention group receive a CD and booklet of relaxation and distraction stories to listen to/read during the preoperative period. Preoperative anxiety is assessed by the child life specialist in the preoperative holding area. Ease of induction and emergence from anesthesia are rated by the anesthesia care provider. Post-hospital behaviors are reported by the parents one week after discharge. It is hypothesized that children receiving the intervention will have less anxiety, easier induction and emergence from anesthesia, and fewer changes in post-hospital behaviors than children in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4-12 years of age scheduled for elective surgery

Exclusion Criteria:

* Children < 4 years of age or > 12 years of age

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2004-02-17 (Actual); Primary Completion 2007-08-16 (Actual); Study Completion 2007-08-16 (Actual)

PRIMARY OUTCOMES:
do children who receive the intervention have less anxiety, easier induction and emergence from anesthesia

SECONDARY OUTCOMES:
do children who receive the intervention have fewer changes in post-hospital behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Joel R Wish, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States